CLINICAL TRIAL: NCT01113229
Title: Combined Use of Oxytocin and Misoprostol in the Prevention of Post Partum Haemorrhage
Acronym: CYTOCINON
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: reason of halt prematurely: futility of the trial
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P 081104; 2009-013177-18 (EudraCT Number)
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Hemorrhage; Complicating Delivery
Keywords: Post Partum Haemorrhage,; oxytocin,; misoprostol,; prevention,; delivery.
MeSH Terms: conditions — Hemorrhage; Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): 10 UI of oxytocin IV during delivery of the anterior shoulder of the newborn and two misoprostol tablets taken orally (400µg) following cord clamp
  Interventions: Drug: Misoprostol
- PLACEBO (Placebo Comparator): 10 UI of oxytocin IV during delivery of the anterior shoulder of the newborn and two placebo tablets taken orally following cord clamp.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — two misoprostol tablets taken orally (400µg)
  Other Names: two misoprostol tablets taken orally (400µg

SUMMARY:
To demonstrate that the combined used of oxytocin and misoprostol prevent from post partum haemorrhage better than oxytocin alone, following vaginal birth at 36 to 42 weeks.

DETAILED DESCRIPTION:
Objective :

To demonstrate that the combined used of oxytocin and misoprostol prevent from post partum haemorrhage better than oxytocin alone, following vaginal birth at 36 to 42 weeks'.

Method :

Double blinded Randomized controlled trial in two centers over 30 months.

Treatment :

Patients will be randomly allocated into one of the two following group :

Group A : 10 UI of oxytocin IV during delivery of the anterior shoulder of the newborn and two misoprostol tablets taken orally (400µg) following cord clamp.

Group B: 10 UI of oxytocin IV during delivery of the anterior shoulder of the newborn and two placebo tablets taken orally following cord clamp.

Number of patients:

1550 patients per group (one third reduction of occurrence with alpha and beta set at 0.05 and 0.20 respectively). Patients were included in the study during 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Women>18 years,
* during first stage of normal labor,
* at 36 to 42 weeks,
* with epidural analgesia and informed signed consent

Exclusion Criteria:

* Cesarean section delivery,
* clotting disorders,
* prostaglandin allergy,
* absent consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1721 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of post partum hemorrhage > 500mL in 1 hour | 1 HOUR

SECONDARY OUTCOMES:
Occurrence of post partum hemorrhage > 1000mL in 1 hour | 1 HOUR

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rozenberg, MD, Principal Investigator — CHI POISSY ST GERMAIN
Locations (1):
- Chi Poissy St Germain, Poissy, France

REFERENCES:
- [Derived] Voillequin S, Quibel T, Rozenberg P, Rousseau A. Duration of the second and third stages of labor and risk of postpartum hemorrhage: a cohort study stratified by parity. BMC Pregnancy Childbirth. 2025 Feb 11;25(1):143. doi: 10.1186/s12884-025-07229-4. PMID 39934771
- [Derived] Quibel T, Ghout I, Goffinet F, Salomon LJ, Fort J, Javoise S, Bussieres L, Aegerter P, Rozenberg P; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Active Management of the Third Stage of Labor With a Combination of Oxytocin and Misoprostol to Prevent Postpartum Hemorrhage: A Randomized Controlled Trial. Obstet Gynecol. 2016 Oct;128(4):805-11. doi: 10.1097/AOG.0000000000001626. PMID 27607864